CLINICAL TRIAL: NCT00490958
Title: Effects Of Telmisartan Added To Angiotensin Converting Enzyme Inhibitors On Mortality And Morbidity In Haemodialysed Patients With Chronic Heart Failure: A Double-Blind Placebo-Controlled Trial
Brief Title: Telmisartan in Haemodialysis Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Campania Luigi Vanvitelli (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tchf-01-01
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Last update posted 2008-10-17 (Estimated); Status verified 2007-11

CONDITIONS: Heart Failure, Congestive
Keywords: heart Failure; haemodialysis; telmisartan; angiotensin converting enzyme inhibitor
MeSH Terms: conditions — Heart Failure | interventions — Telmisartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: telmisartan

SUMMARY:
Background: In haemodialysis patients, chronic heart failure (CHF) is responsible for a high mortality rate but, presently, very little data is available regarding this population.

Aim of the study: Aim of this study was to determine whether telmisartan decreases all-cause and cardiovascular mortality and morbidity in haemodialysis patients with CHF and impaired left ventricular ejection fraction (LVEF) when added to standard therapies with ACE inhibitors.

Methods: A 3-year randomized, double-blind, placebo-controlled, multicentre trial was performed involving 30 Italian clinics. Haemodialysis patients with CHF (NYHA class II and III; LVEF 40%) were randomized to telmisartan or placebo in addition to ACE inhibitor therapy. 332 patients were enrolled (165 telmisartan, 167 placebo), and drug dosage was titrated to a target dose of telmisartan of 80 mg or placebo. Mean follow-up period was 35±5 months. Primary outcomes were all-cause mortality, cardiovascular mortality and CHF hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Adult haemodialysis patients with CHF;
* New York Heart Association (NYHA) class II and III;
* Ejection fraction less or equal to 40% determined within 6 months; and
* Therapy with ACE inhibitors individually optimized and unchanged for 30 days before randomization

Exclusion Criteria:

* Hypotension during dialysis;
* Atrial fibrillation;
* Intolerant to low dose of telmisartan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 1999-01; Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
all cause mortality cardiovascular mortality hospitalization for decompensated heart failure | 36 months

SECONDARY OUTCOMES:
acute non-fatal myocardial infarction | 36 months
combined endpoint (cardiovascular mortality in addition to acute non-fatal myocardial infarction) | 36 months
cardiovascular hospital admission | 36 months
nonfatal stroke | 36 months
coronary revascularization | 36 months
permanent premature treatment withdrawals | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Gennaro Cice, MD, Study Chair — Chair of cardiology Second University of Naples
Locations (1):
- Chair of Cardiology Second University of Naples, Naples, Italy

REFERENCES:
- [Derived] Cice G, Di Benedetto A, D'Isa S, D'Andrea A, Marcelli D, Gatti E, Calabro R. Effects of telmisartan added to Angiotensin-converting enzyme inhibitors on mortality and morbidity in hemodialysis patients with chronic heart failure a double-blind, placebo-controlled trial. J Am Coll Cardiol. 2010 Nov 16;56(21):1701-8. doi: 10.1016/j.jacc.2010.03.105. PMID 21070920